CLINICAL TRIAL: NCT04243772
Title: Metabolic Risk Factors and Stones Composition in Adult Kidney Stone Formers
Status: Completed | Type: Observational
Sponsor: Agnieszka Pozdzik (Other)
Responsible Party: Sponsor-Investigator, Agnieszka Pozdzik, Head of nephrology clinic, Brugmann University Hospital
Organization: Brugmann University Hospital (Other)
Other Study IDs: Metastone study
Record Dates: First submitted 2020-01-24; First posted 2020-01-28 (Actual); Last update posted 2024-04-12 (Actual); Status verified 2024-04

CONDITIONS: Kidney Stone
MeSH Terms: conditions — Kidney Calculi

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Lithiasic patients: Lithiasic patients of the CHU Brugmann Hospital
  Interventions: Other: Data extraction

INTERVENTIONS:
Other: Data extraction — Data extraction from medical files

SUMMARY:
Within the CHU Brugmann hospital, a multidisciplinary Renal Lithiasis and Mineral Metabolism clinic has been inaugurated in 2017. During the first months of 2018, the activities of the clinic have been focalized on the pre-analytical and analytical aspects of metabolic work-up. 15 patients are followed on average per week. The clinic is recognized as one of the 24 core centers of the European Nephrolithiasis Network and it is the only clinic included in this network in Belgium. The actual practice of the clinic has been published in a survey regarding current practice patterns of stone centers across Europe. Following this publication, the members of the board of the European Nephrolithiasis Network have put as common effort to standardize the care of kidney stone formers and obtained endorsement to perform a second survey in each core center. The aim of this initiative is to share information from real patients in aggregate form. Each core center practice will be evaluated by the second survey by an analysis of the robustness of clinical, biological, urological and radiological data.

The main aim of this project consists in the constitution of a clinical, biological, urological and radiological database of followed patients. This database could be shared in aggregate form by using a specialized coding system for the patients. The database will enable the investigators to:

* describe the epidemiological and clinico-biological characteristics of the CHU Brugmann patient population
* gather information about the kidney function outcome
* analyze and classify identified prolithogenics factors
* characterize related metabolic disorders (diabetes mellitus, metabolic syndrome, arterial hypertension, chronic kidney diseases, osteoporosis...)
* identify the patients that could participate in the international trials on kidney stone disease
* identify the patients that will need a specialized genetic testing.
* evaluate the impact of the clinic activity and metabolic work-up on the rate of recurrence of kidney stones in the patient population.

The obtained data will be compared with the global data from the European Nephrolithiasis Network.

DETAILED DESCRIPTION:
Nearly 10% of population suffer from kidney stone disease. Recent review reported that kidney stones represent an underestimated risk factor for further kidney function deterioration, arterial hypertension and cardiovascular diseases. They are furthermore a significant predictor of osteoporotic fractures.

This evidence needs to be very seriously considered in children and adolescent suffering from this disorder. The epidemiological registry data show an alarming, continous increase in the incidence of kidney stones in adults (both sexes) and intriguingly in children. During the last 25 years the incidence of nephrolithiasis in children has increased by approximately 6% to 10% annually and is now 50 per 100 000 adolescents. Stone incidence in children undergoing abdominal imaging more than doubled between 2011 and 2016. Moreover, the changes in stone compositions have been identified and remain relevant pathophysiological aspects in the epidemiology of kidney stones.

Acute nephritic colic access reflects only the end-point of mineral metabolism abnormalities - the kidney stone disease is considered as a chronic, systemic mineral metabolism disorder. The process of kidney stones formation - lithogenesis- is a consequence of imbalance between the promotors and inhibitors in the urine. The patients with kidney stone disease require a complete metabolic assessment.

The three main areas leading to stone formation are metabolism, diet and lifestyle. The main causes of kidney stones are most frequently related to an increase in salt and sugar intake, insufficient water intake and increased incidence of obesity. All this together leads to the supersaturation of several biochemical components excreted physiologically in the urine, resulting in fine in their crystallization, a first step in stone formation.

Metabolic work-up is recommended by the American Urology Association to identify and correct the factors responsible for urinary stone formation such as hypercalciuria, hyperoxaluria, hypocitraturia or abnormalities of urinary pH. The metabolic work-up includes the collection of urine during 24h. This is the most useful test, giving information about the patient's average chemical risk of stone formation and it is the nearest available body fluid to the actual formation and growth of the stone itself. Metabolism is dealt with through a concurrent blood and spot urine test. Diet is handled through a variable method of diary recorded by the patient on his free, home diet. Lifestyle is handled with through a standard questionnaire given by the physician.

Within the CHU Brugmann hospital, a multidisciplinary Renal Lithiasis and Mineral Metabolism clinic has been inaugurated in 2017. During the first months of 2018, the activities of the clinic have been focalized on the pre-analytical and analytical aspects of metabolic work-up. 15 patients are followed on average per week. The clinic is recognized as one of the 24 core centers of the European Nephrolithiasis Network and it is the only clinic included in this network in Belgium. The actual practice of the clinic has been published in a survey regarding current practice patterns of stone centers across Europe. Following this publication, the members of the board of the European Nephrolithiasis Network have put as common effort to standardize the care of kidney stone formers and obtained endorsement to perform a second survey in each core center. The aim of this initiative is to share information from real patients in aggregate form. Each core center practice will be evaluated by the second survey by an analysis of the robustness of clinical, biological, urological and radiological data.

The main aim of this project consists in the constitution of a clinical, biological, urological and radiological database of followed patients. This database could be shared in aggregate form by using a specialized coding system for the patients. The database will enable the investigators to:

* describe the epidemiological and clinico-biological characteristics of the CHU Brugmann patient population
* gather information about the kidney function outcome
* analyze and classify identified prolithogenics factors
* characterize related metabolic disorders (diabetes mellitus, metabolic syndrome, arterial hypertension, chronic kidney diseases, osteoporosis...)
* identify the patients that could participate in the international trials on kidney stone disease
* identify the patients that will need a specialized genetic testing.
* evaluate the impact of the clinic activity and metabolic work-up on the rate of recurrence of kidney stones in the patient population.

The obtained data will be compared with the global data from the European Nephrolithiasis Network.

ELIGIBILITY:
Inclusion Criteria:

* Active or past history of kidney stone (newly diagnosed or with relapse)
* Age and sex matched controls from the hospital

Exclusion Criteria:

- None

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients of the CHU Brugmann Hospital with active or past history of kidney stone (newly diagnosed or with relapse). Medical file data collection starts from 01 January 2018.
Sampling Method: Non-Probability Sample
Enrollment: 350 (Actual)
Dates: Start 2019-11-12 (Actual); Primary Completion 2023-12-12 (Actual); Study Completion 2023-12-12 (Actual)

PRIMARY OUTCOMES:
Urinary tract stone composition | 3 years
  Urinary tract stone composition
Metabolic screen results | 3 years
  Metabolic screen (fasting blood) results
24 hour urine screen results | 3 years
  24 hour urine screen (first basal urine) results

CONTACTS AND LOCATIONS:
Overall Officials: Mohamed El Mallouli, Principal Investigator — CHU Brugmann
Locations (1):
- CHU Brugmann, Brussels, Belgium

IPD SHARING:
Plan to Share IPD: No